CLINICAL TRIAL: NCT06215417
Title: Clinical and Cost Effectiveness of Rotator Cuff Augmentation With Human Dermal Allograft Versus Bovine Collagen Xenograft Patch: a Randomized Controlled Trial
Brief Title: Rotator Cuff Augmentation With Human Dermal Allograft Versus Bovine Collagen Xenograft Patch: A Randomized Controlled Trial
Acronym: HDA v Regen
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB23-0276
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: This study is designed as a parallel group 1:1 randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and research assistants collecting data will be unaware of the treatment assigned until the completion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HDA (Experimental): Human dermal allograft (LifeNet Health Arthroflex graft)
  Interventions: Procedure: Rotator cuff repair
- Regeneten (Active Comparator): Bovine collagen patch xenograft (Smith & Nephew Regeneten)
  Interventions: Procedure: Rotator cuff repair

INTERVENTIONS:
Procedure: Rotator cuff repair — Arthroscopic rotator cuff repair augmented with graft.

SUMMARY:
Randomized controlled trial comparing human dermal allograft with bovine collagen xenograft in rotator cuff repair.

DETAILED DESCRIPTION:
Randomized controlled trial comparing human dermal allograft with bovine collagen xenograft in rotator cuff repair.

Subjects will be randomized intraoperatively after confirmation of inclusion criteria.

Subjects will be followed-up at 3 weeks, 3 months, 6 months, 12 months and 24 months post-operatively.

Primary outcome is Western Ontario Rotator Cuff Index (WORC) at 12 months. Additional outcomes include American Shoulder and Elbow Surgeons questionnaire (ASES), Single Numeric Evaluation (SANE) score, EuroQoL (5 domains) score (a quality of life score), and Visual Analogue Scale, healing rate as determined by Magnetic Resonance Imaging (MRI) scan at 12 months post surgery. To determine the cost utility, data will be collected on the cumulative cost for the total episode of care up to 12 months post surgery inclusive of surgical costs, implant costs, outpatient costs, and medication costs. Quality-Adjusted Life Years (QALYs) gained will be calculated using the mean total cost and the quality of life score (EQ-5D) improvement from pre-operative to 12 months post surgery.

ELIGIBILITY:
Inclusion Criteria:

>18 years

- fully reparable full thickness rotator cuff tear whereby the treating surgeon feels a graft augment is needed to enhance healing

Exclusion Criteria:

* tears where only a partial repair is achieved
* significant glenohumeral joint arthropathy (Hamada grade 2 and above)
* irreparable rotator cuff tears
* patients unable or unwilling to consent or comply with study questionnaires
* patients with upper limb neurological deficits affecting the ipsilateral limb
* workers compensation cases
* cases involving litigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Western Ontario Rotator Cuff Index (WORC) | 12 mos post-op
  rotator cuff quality of life outcome questionnaire

SECONDARY OUTCOMES:
Western Ontario Rotator Cuff Index (WORC) | pre-op, 3 mos, 6 mos, 24 mos post-op
  rotator cuff quality of life outcome questionnaire
Single Assessment Numeric Evaluation (SANE) | pre-op, 3mos, 6mos, 12mos, 24mos post-op
  numeric score indicating shoulder assessment
EuroQOL5D | pre-op, 3mos, 6mos, 12mos, 24mos post-op
  general health assessment score
Shoulder pain assessed by visual analog scale (VAS) | pre-op, 3mos, 6mos, 12mos, 24mos post-op
  assessment of shoulder pain
Anatomic healing | 12mos post-op
  anatomic healing as assessed via MRI

IPD SHARING:
Plan to Share IPD: No
No sharing of IPD.